CLINICAL TRIAL: NCT05531695
Title: A Pilot Study of Moderate Intensity Exercise as Adjuvant Therapy in the Management of Brain and Central Nervous System Cancer
Brief Title: Exercise Study in Brain and CNS Cancer
Acronym: ESIBAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Collaborators: University of Bath (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: R1789
Record Dates: First submitted 2019-02-25; First posted 2022-09-08 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Cancer of Brain and Nervous System
MeSH Terms: conditions — Brain Neoplasms; Neurologic Manifestations | interventions — Exercise; Pliability

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aerobic Exercise (Experimental): Graduated supervised moderate intensity aerobic exercise
  Interventions: Behavioral: Exercise (either aerobic or flexibility)
- Flexibility Exercise (Active Comparator): Home based self-supervised flexibility exercises
  Interventions: Behavioral: Exercise (either aerobic or flexibility)

INTERVENTIONS:
Behavioral: Exercise (either aerobic or flexibility)

SUMMARY:
With a trend for increased survival in patients with Brain and Central Nervous System (CNS) cancers, emphasis is increasingly shifting to improving the quality of life of survivors. Performance status (a quantification tool used in patients with cancer to assess their quality of life and ability to carry out activities of daily living) is a key prognostic factor in Brain and CNS cancers and a good performance status is used in determining whether a patient is offered adjuvant treatment with chemotherapy and radiotherapy following primary surgical treatment. The performance status of a patient is defined by physical and cognitive functioning, and the beneficial effect of aerobic exercise in improving physical functioning (e.g., cardiorespiratory fitness) is well established. Thus, it is anticipated that implementing a supervised moderate intensity aerobic exercise training programme will improve the performance status of patients. An implication of this work is that, exercise regimens could be offered as additional treatment, alongside chemotherapy and radiotherapy, which might increase the chance of survival.

The project design is a randomised controlled trial with two arms in which one group of patients will undergo an aerobic exercise program starting one week before surgery and continuing for three weeks in the post-operative period. Patients enrolled in this trial will continue with standard treatment including neuro-rehabilitation. The control group of patients will be given written instructions on performing flexibility and stretching exercises in addition to their usual care (including neuro-rehabilitation). The primary outcome is performance status as defined by measurements of physical functioning and cognitive ability (e.g., memory, attention, information processing speed). Physical functioning will be assessed by a timed walking test, hand-grip dynamometry and a maximum jump height test. Other measures of well-being will be assessed; including heath related quality of life using the European Quality of Life-5 Dimensions (EQ-5D) and Functional Assessment of Cancer Therapy- Brain (FACT-Br) questionnaires. Secondary outcome measures will be measurements of mood, fatigue and certain biochemical parameters, such as C-reactive protein (CRP), plasma viscosity (PV), full blood count (FBC), uric acid, insulin-like growth factor 1 (IGF-1), and insulin-like growth factor binding protein 3 (IGFBP-3). It is anticipated that a total of 30 patients will be recruited split between the two groups and each participant will not spend more than four weeks in taking part in the study.

DETAILED DESCRIPTION:
Study design:

Randomised controlled trial. Participants will be randomised into one of two groups: intervention or control. Participants in the intervention group will undergo a supervised moderate intensity aerobic exercise programme in addition to routine treatment starting 1 week after their primary treatment (surgery/radiotherapy) for 3 weeks.

Participants in the control group will undergo a programme involving muscle stretching (flexibility) exercises using a combination of active and passive static stretching to target the major muscle tendon units of the neck, shoulder girdle, chest, trunk, lower back, hips, legs (posterior and anterior aspects) and ankles over the same time period as the intervention group. The exercises in this group will be unsupervised. Patients will be provided with written clear instructions listing the stretches to perform. These written instructions will be supplemented with diagrams for each stretch manoeuvre.

Research setting:

The project will be based within the premises of the Hull and East Yorkshire hospital NHS Trust. This is an acute care tertiary centre based over two hospital sites: the Hull Royal Infirmary (HRI) and Castle Hill Hospital (CHH). The neurosurgical ward and operating theatres are based at the HRI site while the inpatient specialist rehabilitation ward and the oncology facilities and clinicians are based at the Queens Centre for Oncology/Haematology within the premises of CHH. The neurosurgery outpatient clinic is also based at CHH site. The facilities and equipment for the exercise intervention will be based in a dedicated specialist inpatient rehabilitation unit on ward 29 at the Queens centre. The Queens Centre is a purpose built oncological facility that co-locates all of the services (including psychology) involved in cancer care apart from surgical services. This protocol and proposal has been utilised in making ethics submission across 2 institutions- the University of Bath and the Hull and East Yorkshire Hospital NHS Trust hosting the study setting.

Demographic information:

Participants' medical history will be obtained from the hospital records. Medical co-morbidities may affect clinical outcome in patients with brain and CNS cancers. However, collected information will be anonymised and patient identification information will remain within the clinical setting. These will be stored under data protection regulations that govern the NHS.

Assessments

There are 3 designated time points in the course of the study during which the assessment tools for the outcome measures will be administered. These are:

1. Baseline. This marks the entry period into the study when informed written consent has been obtained. It is designed to coincide with the first visit to the project base prior to commencing the exercise programme. Fast-track access to neuro-oncology multidisciplinary team assessment clinic within 1-2 weeks of referral is the norm. The nature of this clinical diagnosis is such that surgical intervention in eligible patients is scheduled within 2 weeks of clinic appointment hence the time constraints of the pre-operative phase.
2. The first post-operative assessment. This is scheduled to take place one week after operation in order to allow for tissue healing and post-operative inflammatory processes to settle. It is acknowledged that the post-operative medical stability cannot be predicted and the assessment scheduled for this period may be delayed to such a time when the patient is assessed to be medically stable enough to resume the rehabilitation program. All of this information will be recorded.
3. The final assessment. This will be undertaken following completion of the 3 week exercise programme in the post-operative period. This will also mark the official termination point of the patient intervention part of the study.

ELIGIBILITY:
Inclusion Criteria:

* Adult (aged 18 years plus).
* Diagnosis of a primary brain and CNS cancer.
* Patients with recurrent brain/CNS tumours eligible for further excision surgery will be included. This is because this group of patients are considered to have good performance score and similar in many characteristics to newly diagnosed patients with brain tumour.
* No contraindication to undertaking moderate aerobic physical activity such as unstable angina, acute systemic illness or fever, uncontrolled diabetes, recent embolism (< 4 weeks), resting heart rate > 120 beats per minute, severe uncontrolled hypertension (180/110 mmHg), progressing worsening dyspnoea at rest or exertion over previous 3-5 days and severe anaemia (haemoglobin concentration ≤ 60 g/L).
* Able to provide consent.

Exclusion Criteria:

* Severe ataxia.
* Co-morbidities such as severe cardiovascular or respiratory disease.
* Acute or emergency neurosurgical intervention as primary treatment (the pre-operative exercise phase cannot be implemented).
* Uncontrolled seizure disorder.
* Patients primarily for palliation or on end of life care pathway.
* Patients who require barrier nursing for infection control.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Hand grip strength | 4 weeks
  Hand grip strength in Kg of study participants using portable dynamometry before and after intervention.
6 minute walk test. | 4 weeks
  Distance walked in metres by participants in 6 minutes on a level indoor surface before and after intervention.
Sit and reach test | 4 weeks
  Flexibility measurement in centimetres using a sit and reach box
Vertical jump test | 4 weeks
  Vertical height jumped in centimetres using an electronic jump mat
Karnofsky Performance Status (KPS) | 4 weeks
  Measurement or performace on an ordinal rating scale

SECONDARY OUTCOMES:
Health related quality of life (HRQOL) of participants before and after intervention: questionnaires | 4 weeks
  The HRQOL of patients with primary brain and CNS tumour following primary treatment as measured by the following self-report paper-based questionnaires: These questionnaires will be administered at the three assessment points.
C-reactive protein level | 4 weeks
  C-reactive protein (CRP) in blood samples collected from participants before and after the exercise intervention.
Full Blood Count | 4 weeks
  Full blood count (FBC) as measure of disease burden and inflammatory response
Interleukin-6 assay | 4 weeks
  Interleukin 6 (IL6) in pre and post intervention samples
Plasma viscosity (PV) | 4 weeks
  Plasma viscosity (PV) as a measure of hydration response to exercise intervention.
Insulin-like growth factor 1 (IGF1) | 4 weeks
  Plasma assay of insulin-like growth factor 1 (IGF1) to evaluate metabolic response to intervention.
Insulkin-like Growth Factor Binding Protein -3 (IGFBP3) | 4 weeks
  Serum level of insulin-like growth factor binding protein (IGFBP3) to evaluate the metabolic response to exercise intervention.
Serum Uric acid | 4 weeks
  Serum Uric acid level as a measure of hydration response to exercise intervention will be assessed.
Borg rate of perceived exercition | 4 weeks
  An assessment of individual participants perception of the degree of exertion in relation to their assigned exercise programme using the Borg rating scale of perceived exertion.
Functional independence measure (FIM) and Functional assessment measure (FAM) | 4 weeks
  Measure of functional indepence in performance activities of daily living
Rehabilitation Complexity scale (RCS). | 4 weeks
  Measure of clinical complexity derived from aggegate score of subscales of therapeutic interventions (scored from 0-15)

OTHER OUTCOMES:
Physical activity and exercise readiness questionnaire; physical activity readiness questionnaire (PARQ) | one week
  Exercise readiness and behaviour to be assessed by administering the physical activity readiness questionnaire (PARQ). These are self-report paper based questionnaires which will be administered at baseline only. (Scale of 0-7).
Physical activity and exercise readiness questionnaire: Godin leisure time exercise questionnaire | One Week
  Exercise readiness and behaviour to be assessed by administering the Godin leisure time exercise questionnaire. These are self-report paper based questionnaires which will be administered at baseline only. (Scale 0-99)

CONTACTS AND LOCATIONS:
Overall Officials: James E Turner, PhD, Study Chair — University of Bath
Locations (1):
- Castle Hill Hospital, Hull, East Yorkshire, United Kingdom